CLINICAL TRIAL: NCT05188781
Title: A Phase II Evaluation of Pembrolizumab in Combination With Anlotinib in the Treatment of Refractory or Recurrent High-Grade Serous Ovarian Cancer
Brief Title: Pembrolizumab and Anlotinib in the Treatment of High-Grade Serous Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, zhangxiaochun, Cancer precision Medicine Center, The Affiliated Hospital of Qingdao University
Other Study IDs: HGSOC-001
Record Dates: First submitted 2021-11-29; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: High-Grade Serous Ovarian Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pembrolizumab combined with Anlotinib: Pembrolizumab 200 mg every 3 weeks, Anlotinib 12 mg/day, orally;2weeks treatment followed by 1week off
  Interventions: Drug: Pembrolizumab combined Anlotinib

INTERVENTIONS:
Drug: Pembrolizumab combined Anlotinib — Pembrolizumab 200 mg every 3 weeks, Anlotinib 12 mg/day, orally;2weeks treatment followed by 1week off

SUMMARY:
Primary:

To evaluate improvement in progression-free survival for patients treated with anti-PD1 pembrolizumab in combination with Anlotinib as compared to pembrolizumab single treated Secondary: To obtain pilot data on clinical response rates using both RECIST1.1 criteria (Response Evaluation Criteria in Solid Tumors) and immune related response criteria (irRECIST).

Objectives • To obtain data on changes in tumor microenvironment prior to and subsequent to therapy and, to screen for potential biomarkers to predict clinical benefit combination in the study population.

* To assess the impact of the combination of anlotinib and pembrolizumab
* To determine the safety and tolerability of the treatment of anlotinib and pembrolizumab
* To evaluate overall survival in patients treated with anti-PD-1 pembrolizumab and anlotinib

DETAILED DESCRIPTION:
This is an open label Phase II study of anti-PD1 antibody pembrolizumab, in combination with anlotnib in patients with recurrent platinum sensitive, resistant or refractory. The study will enroll approximately 40 evaluable patients in total. Accrual is expected to take 18 months.

Disease Evaluation: CT at Baseline, after 3rd cycle, after 6th cycle then, after every 6th cycle (or sooner if disease progression) Adverse Events: Day 1 of each cycle, end of treatment, safety follow-up.

Hematology: Baseline, Day 1 of each cycle, end of treatment, safety follow-up . Chemistry: Baseline, Day 1 of each cycle, end of treatment, safety follow-up Performance Status: Baseline, Day 1 of each cycle, end of treatment, post treatment evaluations Full Physical Examination (including basic neurological examination, vital signs, and body weight): Baseline, Day 1 Cycle 1, Day 1 of every 3rd cycle, end of treatment, post treatment evaluations Directed Physical Examination (including basic neurological exam, vital signs, and body weight): On cycles not requiring a full physical examination (e.g. cycles 2 and 3, cycles 5 and 6) Vital Signs: Baseline, Day 1 of each cycle, end of treatment evaluations Pregnancy test: Within 72 hours prior to receiving first dose of study treatment in patients of childbearing potential post treatment PT/INR and APTT: Baseline, Cycle 6 Day 1, Cycle 12 Day 1, end of treatment, safety follow-up.

Urinalysis: Baseline, Cycle 1Day 1, every 2nd cycle after Cycle 1, end of treatment.

UPCR Ratio: Baseline, Cycle 1Day 1 and, Day 1 of every 2nd cycle. T3, FT4, and TSH: Baseline, Cycle 3 Day 1 then Day 1 of every 3rd cycle, end of treatment, safety follow-up Tissue Biopsy: Baseline, 2-3 weeks after Cycle 3, end of treatment (optional) Blood Collection (correlative studies): Baseline (within 2 weeks prior to treatment initiation), Cycle 2 - Day 1, Cycle 4- Day 1, Cycle 7- Day 1, Cycle 10 -Day 1, and at the end of study treatment or at time of discontinuation (within two weeks after the last treatment cycle is completed) or, at the time of disease progression or for any other reason that requires study treatment termination, whichever occurs sooner. On those patients, who have already completed 10 cycles, the one additional correlative blood sample will be collected at the time of their next cycle.

Safety Analysis: The frequency of toxicities will be tabulated by grade across all dose levels and cycles. Toxicity rates will be estimated using 90% confidence intervals, which will be obtained using Jeffreys prior method. All participants who receive any study treatment will be considered evaluable for toxicity. The overall and progression free survival will be summarized using standard Kaplan-Meier methods, with estimates of median survival and given survival rates will be obtained with 90% confidence intervals.

Efficacy Analysis: The overall and progression free survival will be summarized using standard Kaplan-Meier methods, with estimates of median survival and given survival rates will be obtained with 90% confidence intervals. Objective tumor response will be tabulated for all patients that completed at least three cycles of the proposed treatment Correlative Data Analysis: The blood and tumor samples will be collected as biomarkers and will be reported using the appropriate descriptive statistics depending on clinical outcome. Associations between these markers and PFS will be evaluated using Cox regression models; while associations with tumor response will be evaluated using logistic regression models.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, participants must meet the following criteria:

Age more than 18 years of age on day of signing informed consent. Have an ECOG Performance Status of 0 or 1 (refer to Appendix A). Have measurable disease per RECIST 1.1 or irRECIST criteria present. Participant may have serous, endometrioid, clear cell, mucinous or undifferentiated type of recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer.

Histologic confirmation of the original primary tumor is required via the pathology report.

Participant can be either platinum-sensitive (platinum free interval (PFI) ≥ 6 months prior to recent recurrence) or platinum-resistant (PFI < 6 months prior to recent recurrence). If the participant has a platinum sensitive disease, she may only enroll in this clinical trial if there is a contraindication for her to receive further treatment with platinum-based chemotherapy (such as serious persistent toxicity or severe hypersensitivity to platinum agents or she declines standard of care).

Participant must be willing to undergo core or excisional biopsy of a tumor lesion within 4 weeks (28 days) prior to initiation of treatment on Day 1and, after 3 cycles of study treatment.

Participants for whom newly obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Principal Investigator.

Have the following clinical laboratory values:

Absolute neutrophil count (ANC): ≥ 1,500 /mcL Platelets: ≥ 100,000 / mcL Hemoglobin: ≥ 9 g/dL or 5.6 mmol/L without transfusion or EPO dependency(within 7 days of assessment) Serum creatinine: ≤1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance ≥ 60 mL/min for participant with creatinine levels > 1.5 institutional ULN (refer to Appendix B). GFR can also be used in place of creatinine or CrCl.

Urine Protein Creatine Ratio (UPCR) < 1 prior to enrollment Serum total bilirubin: ≤ 1.5 X ULN OR direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT): ≤ 2.5 X ULN OR ≤ 5 X ULN for participants with liver metastases Albumin: > 2.5 mg/dL International Normalized Ratio (INR) or Prothrombin Time (PT): ≤1.5 unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants Activated Partial Thromboplastin Time (aPTT): ≤1.5 X ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants Participants of childbearing potential must have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Participants of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year). Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.

Participant has recovered from toxicities of prior chemotherapy or other therapy (to grade 2 or less).

Participant may have received prior investigational therapy (including immune therapy). Participant may have received prior hormonal therapy.

Participant may have received anlotinib in the past. Participant has had at least 4 weeks of postoperative recovery from surgery prior to enrollment to ensure complete wound healing. Participants with bowel resections at surgery should begin protocol at least 42 days after surgery.

Ability to swallow and retain oral medication. Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

Participants will be excluded from this study for the following:

Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.

Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment or, is taking any other medication that might affect immune function.

Has a known history of active TB (Bacillus Tuberculosis). Hypersensitivity to bevacizumab, cyclophosphamide, pembrolizumab or any of its excipients.

Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.

Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

Note: Participants with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy and, has to be at least 28 days after the surgery Has a known additional malignancy that is progressing or requires active treatment: exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or cervical cancer in situ that has undergone potentially curative therapy.

Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.

Has active autoimmune disease that has required systemic treatment in the past 6 months (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.

Has known history of, or any evidence of active, non-infectious pneumonitis. Has an active infection requiring systemic therapy. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Is pregnant or breastfeeding or expecting to conceive within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.

Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies). Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).

Has received a live vaccine within 30 days of planned start of study therapy.

o Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Active or history of inflammatory bowel disease (colitis, Crohn's), diverticulitis, irritable bowel disease, celiac disease, or other serious, chronic, gastrointestinal conditions associated with diarrhea. Active or history of systemic lupus erythematosus or Wegener's granulomatosis.

Participant has clinical symptoms or signs of partial or complete gastrointestinal obstruction or, requires parenteral hydration and/or nutrition.

Participant requires, or is likely to require, more than a two - week course of corticosteroids for intercurrent illness. Participant must complete the course of corticosteroids 2 weeks before screening to meet eligibility.

Participant has a serious, non- healing wound, ulcer, or bone fracture.

Participant has a clinically significant cardiovascular disease including:

Uncontrolled hypertension, defined as systolic > 150 mmHg or diastolic > 90 mmHg Myocardial infarction or unstable angina within 6 months prior to enrollment New York Heart Association (NYHA) Grade II or greater congestive heart failure (refer to Appendix F) Participant has a grade II or greater peripheral vascular disease Participant has a clinically significant peripheral artery disease (e.g. those with claudication, within 6 months) Participant has organ allografts. Participant is receiving medication(s) that might affect immune function. Unwilling or unable to follow protocol requirements.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The study will enroll approximately 40 evaluable patients in total (includes a safety lead-in cohort of n=5). Accrual is expected to take 18 months.
  Study treatment is for 12 months (or a maximum of 17 cycles), with a follow-up period of up to 3 years from initiation of study treatment; for a total study duration of approximately 5 years.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
ORR | 01.01.2019 to 01.01.2022
  objective response rate

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaochun Zhang, Qingdao, Shandong, China